CLINICAL TRIAL: NCT07086131
Title: Impact Of Adding Inspiratory Muscle Training To Cardiac Rehabilitation On Exercise Responses In Heart Failure
Brief Title: A Study Investigating the Impact of IMT With CR On Exercise Responses In HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joshua R. Smith, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 25-005871; 1R01HL176491-01 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Inspiratory muscle training (IMT) (Experimental): IMT performed at 40% maximal inspiratory pressure (MIP) for 30 minutes 3 days a week for 12 weeks.
  Interventions: Device: Powerbreathe
- SHAM (Sham Comparator): IMT performed at 5% maximal inspiratory pressure (MIP) for 30 minutes 3 days a week for 12 weeks.
  Interventions: Device: Powerbreathe

INTERVENTIONS:
Device: Powerbreathe — The breathing training will consist of using the PowerBreathe for 12 weeks. The PowerBreathe is an inspiratory pressure threshold trainer. The valve blocks the airflow until the threshold pressure is achieved by breathing in forcefully into the device.

SUMMARY:
The purpose of this study is to compare the impact of inspiratory muscle training (IMT) combined with cardiac rehabilitation (CR) on cardiovascular function in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria

HFrEF Patients: (≥18 yrs) receiving guideline directed pharmacologic medical therapy for >6 weeks (those with contraindications to medical therapy will meet inclusion criteria), NYHA symptoms I-III, no hospitalizations in the >3 months, have a body mass index ≤45 kg/m2, currently be non-smokers with <30 pack year history and be able to exercise (i.e. without significant orthopedic limitations or musculoskeletal disorders limiting their ability to exercise).

Exclusion Criteria

1. sustained ventricular tachycardia and/or ventricular fibrillation within 21 days of visit 1;
2. second or third degree heart block;
3. body mass index >45 kg/m2;
4. current smokers and/or smoking history >30 pack years;
5. pregnant women (testing will be done by research team if requested);
6. glomerular filtration rate of <30 mL/min/1.73m2 (initial screen via clinical record within the past 6 months and this will be assessed on Visit 1);
7. individuals who are not able to engage in exercise;
8. symptomatic peripheral artery disease;
9. asthmatic patients with a low symptom perception and suffer frequency, severe exacerbations or with an abnormally low perception of dyspnea;
10. ruptured eardrum or any other condition of the ear;
11. history of spontaneous pneumothorax or osteoporosis with a history of rib fractures;
12. history of lung disease.

For individuals agreeing to undergo dual energy x-ray absorptiometry (DEXA) scanning for measurement of body composition as part of their study visit, additional exclusion criteria apply: recently administered gastrointestinal contrast or radionuclides; severe degenerative changes or fracture deformity in measurement areas; or inability to attain correct position and/or remain motionless for the measurement period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in locomotor muscle blood flow during exercise | Baseline, 12 weeks
  Locomotor muscle blood flows will be measured via Doppler-ultrasound. This will be measured in mL/min.
Change in respiratory muscle cost of breathing (VO2) | Baseline, 12 weeks
  Respiratory muscle cost of breathing is the oxygen uptake (VO2) to the respiratory muscles. Respiratory muscle VO2 is expressed as milliliters of oxygen per kilogram of body mass per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Smith, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No